CLINICAL TRIAL: NCT00893945
Title: A Phase I Study of Autologous Dendritic Cells Pulsed With Autologous Apoptotic Tumor Cells (DC/AAT) Administered Intradermally to Cancer Patients With Brain Tumors
Brief Title: Autologous Dendritic Cells Pulsed With Autologous Apoptotic Tumor Cells Administered to Patients With Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RDA-0611
Record Dates: First submitted 2008-12-05; First posted 2009-05-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC/AAT vaccine (Experimental): Intradermal injection of 3 Autologous dendritic cell vaccines (DC/AAT, DC/AAT-flu, DC/KLH) that have been co-cultured with autologous apoptotic tumor specimens.
  Interventions: Drug: DC/AAT; Drug: DC/AAT-Flu; Drug: DC/KLH

INTERVENTIONS:
Drug: DC/AAT — Autologous dendritic cells that have been co-cultured with autologous apoptotic tumor (AAT) specimens.
  Other Names: Dendritic cell/autologous apoptotic tumor
Drug: DC/AAT-Flu — Intradermal injection of Autologous dendritic cell vaccine (DC/AAT-Flu) after co-culture with flu-infected AAT
  Other Names: dendritic cell/flu-infected autologous apoptotic tumor
Drug: DC/KLH — Intradermal injection of Autologous dendritic cell vaccine (DC/KLH) which have been co-cultured with Keyhole pimpit hemocyanin (KLH) as a positive control.
  Other Names: dendritic cell/Keyhole Limplet hemocyanin

SUMMARY:
This study involves cancer research and the purpose is to assess the safety and activity of a type of vaccine as immune therapy for cancer.

This vaccine will be made from each participant's own immune cells (called dendritic cells) obtained by blood donation. Dendritic cells (DCs) are immune cells whose role is to identify foreign material in the body (such as bacteria, viruses, or tumor cells).

When DCs recognize this material, they use it to activate other cells of the immune system to mount an attack against that foreign material. In the Laboratory of Molecular Neuro-Oncology, each participant's DCs will be loaded with samples of their own tumor cells that were obtained at surgical resection. These tumor cells are killed in the laboratory using a special protocol, and then "fed" to the DCs. The DCs "eat" this material, and these "fed" DCs make up the vaccine.

DETAILED DESCRIPTION:
If you are eligible, and you decide to join this research study, you will get two to three shots of the experimental vaccine, each three weeks apart.

You will then have a follow up period where we will monitor you and your medical records for any affects of the experimental treatment.

ELIGIBILITY:
Inclusion Criteria:

Screening to determine eligibility (with the exception of HLA haplotyping) will be completed within 45 days fo study entry.

1. Disease Characteristics

   Histologically confirmed brain cancers, reviewed at MSKCC. Pathologic examination will be of surgical resection specimens deemed of suitable quality for definitive diagnosis by the histopathologist.

   Primary Brain Tumors:
   * Anaplastic astrocytoma
   * Glioblastoma multiforme
   * Anaplastic oligodendroglioma
   * Malignant mixed oligoastrocytoma

   Secondary (metastatic) brain tumors - newly diagnosed or recurrent disease
   * All histological grade of disease accepted

   Surgically accessible tumor for which resection is indicated. Tumors may be from initial resections or re-resections. Recovery of a minimum of 1x10^7 tumor cells ex vivo is required.

   Patients with primary brain tumors must have been previously treated with conventional therapy.
2. Prior/Concurrent Therapy

   1. Recovered from toxicity of any prior therapy
   2. Biologic Therapy

      * No concurrent other immunotherapy and no prior immunotherapy with any of the components of the current regimen (autologous DCs, cancer cells, or KLH)
   3. Chemotherapy:

      * No concurrent immunomodulatory or chemotherapy therapy
      * Chemotherapy, including temozolomide and local chemotherapies such as Gliadel Wafers, must be deferred until after last post-vaccine leukapheresis
   4. Endocrine evaluation/therapy:

      * steroid dose no greater than 1mg daily dexamethasone (or equivalent)
   5. Radiotherapy:

      * No concurrent brain radiation
   6. Surgery:

      * Surgical resection must have been completed independently of this study, and suitable samples obtained for vaccine production
3. Patient Characteristics

   1. Age: 18 and over, able to give written informed consent. May be obtained through use of legal representation such as a health care proxy
   2. Performance status: Karnofsky 60-100%
   3. Life expectancy: at least 4-6 months
   4. Hematopoietic:

      * WBC greater than 3,800
      * Absolute lymphocytes greater than 500
      * Absolute neutrophil counter great than 1,500/mm^3
      * Platelets greater than 100,000/mm^3
      * Hb greater than or equal to 10g/dL
   5. Hepatic: bilirubin less than 2mg/dL OR SGOT less than 2x ULN
   6. Renal: Creatinine no greater than 2mg/dL
   7. Cardiovascular:

      * No NYHA class III/IV status
      * No active angina, uncontrolled clinically significant cardiac arrythmia, recent (6 months) myocardial infarction
   8. Pulmonary: No symptomatic pulmonary disease or pulse oximetry less than 93% on room air
   9. Endocrine: No history of autoimmune thyroid disease
   10. Radiographic: baseline contrast-enhanced MRI or CT scan of brain post surgical resection
   11. Coagulation: No unexplained INR >2

Exclusion criteria:

* No active infection requiring antibiotics
* No history of HIV, hepatitis B or hepatitis C virus infection, no history of high risk behavior for such infection (intravenous drug abuse, men having unprotected sex with men). Laboratory evaluation for HIV, hepatitis B, hepatitis C to be obtained prior to study entry
* No history of hypersensitivity to vaccine components
* No history of autoimmune or vasculitic disease (including but not limited to systemic lupus erythematosis, Hashimoto's thyroiditis, rheumatoid arthritis, systemic necrotizing vasculitides (polyarteritis nodosa group), hypersensitivity vasculitis, Wegener's granulomatosis), scleroderma, multiple sclerosis, juvenile-onset insulin-dependent diabetes
* No medical or psychiatric illness or social condition that, in the opinion of the investigator, would interfere with adherence to study requirements
* No alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Toxicity- assessment of safety and tolerability | week 0 to week 9

SECONDARY OUTCOMES:
Measurable disease | baseline and after completion of vaccination
Activity-monitoring both clinical and immunologic parameters | week 0 to week 9

CONTACTS AND LOCATIONS:
Overall Officials: Robert Darnell, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- [Derived] Frank MO, Kaufman J, Parveen S, Blachere NE, Orange DE, Darnell RB. Dendritic cell vaccines containing lymphocytes produce improved immunogenicity in patients with cancer. J Transl Med. 2014 Dec 5;12:338. doi: 10.1186/s12967-014-0338-3. PMID 25475068